CLINICAL TRIAL: NCT03813121
Title: The Effects of Sedatives on Tobacco Use Disorder
Acronym: SED-TUD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB000229077
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-08

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- midazolam intravenous infusion (Experimental): single midazolam infusion (0.02 mg/kg over 20 minutes)
  Interventions: Drug: midazolam intravenous infusion
- placebo intravenous infusion (Placebo Comparator): single placebo infusion (saline over 20 minutes)
  Interventions: Drug: placebo intravenous infusion
- ketamine intravenous infusion (Experimental): single ketamine infusion (0.5 mg/kg over 20 minutes)
  Interventions: Drug: ketamine intravenous infusion

INTERVENTIONS:
Drug: midazolam intravenous infusion — Participants will receive a single drug infusion
  Arms: midazolam intravenous infusion
Drug: placebo intravenous infusion — Participants will receive a single placebo infusion
  Arms: placebo intravenous infusion
Drug: ketamine intravenous infusion — Participants will receive a single drug infusion
  Arms: ketamine intravenous infusion

SUMMARY:
This proposal will obtain preliminary data on the effect of a single sub-anesthetic dose of a sedative on cigarette craving and smoking behavior as well as measuring tolerability and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* smoke at least 5 cigarettes per day
* smoked at least 2 years
* negative urine drug screen for psychoactive drugs and negative breath alcohol concentration
* live in Little Rock AR or surrounding area

Exclusion Criteria:

* unstable or stable medical condition that would interact with study medication or participation
* serious head trauma or neurological disorder
* hypertension, abnormal ECG or metabolic blood results
* meet criteria for psychosis, schizophrenia, major depressive disorder, or bipolar disorder
* use of psychoactive drugs or medications
* BMI > 40
* among women, pregnancy or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merideth Addicott, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants must be screened for eligibility before being assigned to a group. Participants deemed ineligible were excluded from the study.
Period: Overall Study
Arm/Group | Placebo Intravenous Infusion | Ketamine Intravenous Infusion
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Intravenous Infusion | Ketamine Intravenous Infusion | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.2) | 35.5 (15.4) | 36.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Side Effects
Description: drug side effects scale: severity scale from 1 (not at all) to 7 (extremely) for symptoms of nausea, dizziness, sleepiness, strange thoughts, hallucinations, confusion, anxiousness, and headache. The average score across all side effects is reported.
Time Frame: about 1 week post infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Intravenous Infusion | Ketamine Intravenous Infusion
Number analyzed (Participants) | 4 | 6
score on a scale | 1.3 (0.2) | 1.4 (0.7)

ADVERSE EVENTS:
Time Frame: For 7 days post drug administration.
Arm/Group | Placebo Intravenous Infusion | Ketamine Intravenous Infusion
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 1/4 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Intravenous Infusion (N=4) | Ketamine Intravenous Infusion (N=6)
Nausea (General disorders) | 0 (0) | 1 (1)
Emotional distress (General disorders) | 0 (0) | 1 (1)
motor incoordination (General disorders) | 0 (0) | 1 (1)
Tingling (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The planned enrollment was 12 people. Investigator decided to complete the study early at 10 people because the principal investigator was leaving the institution and the logistics of running this remotely were too difficult. The last participant's last visit occurred, no new subjects were enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT03813121/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT03813121/ICF_001.pdf